CLINICAL TRIAL: NCT07120009
Title: Selective Caries Removal Versus Partial Pulpotomy in the Treatment of Deep Caries: A Randomized Controlled Trial
Brief Title: Partial Pulpotomy vs Selective Removing in Deep Caries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, zeliha gonca bek kurklu, associate professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: cu dişhekimligi
Record Dates: First submitted 2025-06-24; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Deep Dentin Caries in Mature Permanent Teeth
Keywords: Vital pulp therapy; Deep caries; Selective caries removal; Partial pulpotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- selective caries removal (Experimental): Deep caries lesions will be treated with selective caries removal and followed up
  Interventions: Procedure: selective caries removal
- partial pulpotomy (Experimental): Deep caries lesions will be treated with partial pulpotomy and followed up
  Interventions: Procedure: partial pulpotpmy

INTERVENTIONS:
Procedure: selective caries removal — The caries is not completely removed but covered with a remineralizing material. Its purpose is to maintain pulp vitality.
  Arms: selective caries removal
Procedure: partial pulpotpmy — Complete cleaning of the caries resulting in pulp expose. pulp tissue is surgically removed by 1-3 mm.The aim is to remove the inflamed superficial pulp tissue to allow healing from the underlying healthy tissue.
  Arms: partial pulpotomy

SUMMARY:
The aim of this study was to compare the one-year results of selective caries removal and partial pulpotomy treatments in terms of pulp survival and the need for further endodontic treatment in deep carious lesions.Individuals aged 18-65 years with medically healthy mature permanent teeth with deep caries will be included. The included teeth will be randomly assigned to the selective caries removal or partial pulpotomy group. Follow-up evaluations will be performed at 6 months and 12 months. The main outcome is pulp survival as determined by clinical and radiographic success.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65
* ASA I or II general health status
* Deep primary or secondary caries lesion (up to 75% dentin thickness)
* Restorable permanent teeth with mature apex
* Teeth without clinical and radiographic periapical pathology

Exclusion Criteria:

* Pregnancy
* Periapical lesion
* Spontaneous pain or tenderness to palpation
* Teeth for which pulp opening or crown/root supported prosthesis is planned
* Localized severe periodontitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain | 6th and 12th month
  Detailed medical history
  * Is the pain constant or intermittent?
  * How severe is the pain? The outcome will be evaluated using the Visual Analog Scale (VAS), which ranges from 0 to 10, with higher scores indicating a worse outcome.
Periapical pathology | 6th and 12th month
  Standardized digital periapical radiographs will be taken using the long cone paralleling technique to assess periapical status, presence of radiolucent lesions, and periodontal ligament space. Radiographs will be obtained at baseline, 6 months, and 12 months to monitor treatment outcomes and detect any pathological changes.
Tenderness to percussion | 12th month
  1. Usually, the back of a dental mirror handle or the handle of a periodontal probe is used.
  2. First, vertical percussion (lightly tapping the occlusal surface from above) is performed, followed by lateral percussion (lightly tapping the side of the tooth) if necessary.
  3. It is compared with other teeth in the same area. If the pain is only in one tooth, it suggests pathology.
  4. The patient describes the pain as "aching," "discomfort," or "severe pain." This severity indicates the severity of the inflamation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chua SKX, Sim YF, Wang WC, Mok BYY, Yu VSH. One-year outcome of selective caries removal versus pulpotomy treatment of deep caries: A pilot randomized controlled trial. Int Endod J. 2023 Dec;56(12):1459-1474. doi: 10.1111/iej.13978. Epub 2023 Oct 5. PMID 37795835